CLINICAL TRIAL: NCT07147855
Title: Take Your Sexuality Back - a Feasibility Study of a New Intervention for Sexually Traumatized Women: Preliminary Evaluations of Efficacy and Outcome Measurements
Brief Title: A Feasibility Mixed Methods Study of the Intervention Take Your Sexuality Back for Sexually Traumatized Women.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: University of Agder (Other); NTNU Health (sponsor) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REK829297
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Posttraumatic Stress Symptoms; Sexual Abuse; Sexual Trauma
MeSH Terms: conditions — Sexual Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group "Take your sexuality back" (Experimental): A 12 week group intervention
  Interventions: Behavioral: Take your sexuality back

INTERVENTIONS:
Behavioral: Take your sexuality back — A 12 weeks group program.

SUMMARY:
This study looks at the potential effects of a new group treatment called "Take Your Sexuality Back", designed for women who have experienced sexual trauma. Investigators will collect information in two ways-through forms that participants fill out themselves and through ECG measurements during a stress tests. Data will be collected before the treatment, right after it, and again three months later. When all data are collected and analyzed investigators will carry out in-depth interviews with participants and explore how they felt about being tested and how they understand the results -especially if some numbers look unusual or surprising. The goal with this study is to create a strong foundation for a future larger-scale study of the treatment by testing the methods, estimating the size of possible effects and identify outcome measurements that are experienced as meaningful to the participants.

ELIGIBILITY:
Inclusion Criteria:

1. A history of sexual trauma.
2. Experience trauma-related sexual problems.
3. Age between 18 and 65 years.
4. Enough competence in Norwegian to participate in a psychoeducational group.

Exclusion Criteria:

1. Acute suicidality.
2. Serious substance abuse interfering with treatment
3. Severe dissociative or psychotic disorders.
4. Current life crisis interfering with treatment.
5. Living in an abusive relationship. -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
PTSD-symptoms and complex PTSD symptoms | From enrollment to 3 month after end of treatment (12 weeks treatment)
  The international trauma questionnaire (ITQ). Zero (0) is equivalent to nothing and 4 indicates extremely. Higher scores mean worse outcome.
Sexual satisfaction | From enrollment to 3 months after end of treatment (12 weeks intervention)
  The Sexual Satisfaction Scale for women (SSS-W). Different Likert scales. Higher scores mean worse outcome. Higher scores mean better outcome.
Sexual shame | From enrollment to 3 months after end of treatment (12 weeks intervention).
  The Sexual shame index-revised (SSI-R). One (1) is equivalent to strongly disagree and 6 indicates strongly agree. Higher scores mean worse outcome.
Interoceptive awareness | From enrollment to 3 months after end of treatment (12 weeks intervention).
  The Multidimensional Assessment of Interoceptive Awareness (MAYA 2). Zero is equivalent with never and 5 indicates always. Higher scores mean better outcome.
Responses to script-driven imagery. | From enrollment to 3 months after end of treatment (12 weeks intervention).
  The Responses to script-driven imagery (RSDI) measures emotional, cognitive, and physiological responses in the script-driven imagery procedure. Zero is equivalent to "not at all" and six (6) indicates "very much". Higher scores mean worse outcome.
Touch body map | From enrollment to 3 months after end of the treatment (12 weeks intervention).
  Touch Body Map is an instrument for mapping how the body reacts to touch. Participants color the outlines of a human figure with three colors to mark how different areas of the body react to touch form a loved one. The body map gives a non-verbal expression of how trauma is embodied. The percentage of the different colors will be calculated to assess possible changes through the process
Change in HRV and SampEn from pre-post and at follow up efter 3 month. | Enrollment to 3 months after end of treatment (12 weeks intervention).
  Cardiovascular measurement (ECG) recorded during a script-driven imagery (SDI). HRV and SampEn.
Participants experiences of being tested and their understanding of the results. | Three month after end of treatment, when all quantitative results are analyzed and calculated.
  In-depth interviews with focus on participants own experiences and understanding og the quantitative results.

CONTACTS AND LOCATIONS:
Overall Officials: Hege Kersten, PhD, Study Director — Research and Innovation Manager
Locations (1):
- Sykehuset Telemark HF, Skien, Norway

IPD SHARING:
Plan to Share IPD: No
Data are sensitive and participants' anonymity cannot be guaranteed.

DOCUMENTS (1):
  • Study Protocol (2025-03-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT07147855/Prot_000.pdf